CLINICAL TRIAL: NCT04800822
Title: A PHASE 1, OPEN-LABEL, MULTI-CENTER, DOSE ESCALATION AND DOSE EXPANSION STUDY TO EVALUATE THE SAFETY, TOLERABILITY, PHARMACOKINETICS, AND PRELIMINARY EVIDENCE OF ANTI-TUMOR ACTIVITY OF PF-07284892 (ARRY-558) AS A SINGLE AGENT AND IN COMBINATION THERAPY IN PARTICIPANTS WITH ADVANCED SOLID TUMORS
Brief Title: PF-07284892 in Participants With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was prematurely discontinued due to strategic reasons. The PF-07284892 program will continue
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C4481001; 2022-502431-18-00 (Registry Identifier: CTIS (EU)); 2022-003166-21 (EudraCT Number); SHP2 (Other: Alias Study Number)
Record Dates: First submitted 2021-03-09; First posted 2021-03-16 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Solid Tumor
Keywords: colorectal cancer; non-small cell lung cancer; B-type Raf proto-oncogene (BRAF) mutation; Ras mutation; anaplastic lymphoma kinase (ALK)-positive; neurofibromatosis type 1 (NF1); ROS1
MeSH Terms: conditions — Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung; Hereditary Sensory and Autonomic Neuropathies; Neurofibromatosis 1 | interventions — lorlatinib; binimetinib; Cetuximab; encorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- PF-07284892 monotherapy (Experimental): Monotherapy dose escalation of PF-07284892 in participants with ALK- or ROS1-positive non-small cell lung cancer (NSCLC), B-type Raf proto-oncogene V600E mutation colorectal cancer (CRC), or RAS- mutant, NF1-mutant or BRAF class 3-mutant solid tumors
  Interventions: Drug: PF-07284892
- PF-07284892 in combination with lorlatinib (Part 2) (Experimental): Combination dose escalation of PF-07284892 in combination with lorlatinib in participants with ALK- or ROS1-positive NSCLC
  Interventions: Drug: PF-07284892; Drug: lorlatinib
- Expansion Phase (Cohort 1) (Experimental): PF-07284892 + lorlatinib in participants with ALK+ NSCLC with prior lorlatinib
  Interventions: Drug: PF-07284892; Drug: lorlatinib
- Expansion Phase (Cohort 2) (Experimental): PF-07284892 + lorlatinib in participants with ALK+ NSCLC with no prior lorlatinib
  Interventions: Drug: PF-07284892; Drug: lorlatinib
- Expansion Phase (Cohort 3) (Experimental): PF-07284892 + encorafenib + cetuximab in participants with BRAF V600E mutant CRC with prior BRAF inhibitor (BRAFi) plus epidermal growth factor receptor inhibitor (EGFRi)
  Interventions: Drug: PF-07284892; Biological: cetuximab; Drug: encorafenib
- Expansion Phase (Cohort 4) (Experimental): PF-07284892 + encorafenib + cetuximab in participants with BRAF V600E mutant CRC with no prior BRAFi plus EGFRi
  Interventions: Drug: PF-07284892; Biological: cetuximab; Drug: encorafenib
- Expansion Phase (Cohort 5) (Experimental): PF-07284892 + binimetinib in participants with RAS- mutant, NF1-mutant or BRAF class 3 mutant solid tumors who have received prior standard of care (SOC)
  Interventions: Drug: PF-07284892; Drug: binimetinib
- PF-07284892 in combination with encorafenib and cetuximab (Part 2) (Experimental): Combination dose escalation of PF-07284892 in combination with encorafenib and cetuximab in participants with BRAF V600E mutant CRC
  Interventions: Drug: PF-07284892; Biological: cetuximab; Drug: encorafenib
- PF-07284892 in combination with binimetinib (Part 2) (Experimental): Combination dose escalation of PF-07284892 in combination with binimetinib in participants with Ras-mutant, NF-1 mutant or BRAF class 3 -mutant solid tumors
  Interventions: Drug: PF-07284892; Drug: binimetinib

INTERVENTIONS:
Drug: PF-07284892 — PF-07284892
  Other Names: ARRY-558
Drug: lorlatinib — lorlatinib
  Other Names: Lorbrena; PF-06463922, Lorviqua
  Arms: Expansion Phase (Cohort 1); Expansion Phase (Cohort 2); PF-07284892 in combination with lorlatinib (Part 2)
Drug: binimetinib — binimetinib
  Other Names: Mektovi, PF-06811462, MEK162
  Arms: Expansion Phase (Cohort 5); PF-07284892 in combination with binimetinib (Part 2)
Biological: cetuximab — cetuximab
  Other Names: Erbitux
  Arms: Expansion Phase (Cohort 3); Expansion Phase (Cohort 4); PF-07284892 in combination with encorafenib and cetuximab (Part 2)
Drug: encorafenib — encorafenib
  Other Names: Braftovi, PF-07263896, LGX818
  Arms: Expansion Phase (Cohort 3); Expansion Phase (Cohort 4); PF-07284892 in combination with encorafenib and cetuximab (Part 2)

SUMMARY:
The purpose of this first-in-patient, open label study is to determine the maximum tolerated dose and/or recommended dose for further study of PF-07284892 as a single agent and in combination with lorlatinib, encorafenib and cetuximab, or binimetinib and evaluate the pharmacokinetics, safety, and preliminary clinical activity of single agent and each combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years at the time of informed consent
* Histological or cytological diagnosis of ALK-positive advanced NSCLC, CRC with BRAF V600E mutation, or RAS- mutant, NF1-mutant or BRAF class 3 mutant solid tumor. Participants with ROS-positive NSCLC are also eligible for Part 1 and 2 (Other ROS1-positive solid tumors may be considered after discussion with the sponsor).
* Documentation evidence of biomarker mutation status
* Part 3:

ALK-positive NSCLC with prior lorlatinib and no prior platinum-based chemotherapy (Cohort 1); with prior lorlatinib and prior platinum-based chemotherapy (Cohort 2); or with no prior lorlatinib (Cohort 3).

BRAF V600E mutant CRC participants resistant to BRAFi plus EGFRi (Cohort 4 ); refractory to BRAFi plus EGFRi (Cohort 5); or BRAFi plus EGFRi naïve (Cohort 6).

RAS- mutant, NF1-mutant or BRAF class 3 mutant solid tumors who have received prior SOC (Cohort 7).

Exclusion Criteria:

* Brain metastasis larger than 4 cm
* Active malignancy within 3 years
* Systemic anti-cancer therapy or small molecule therapeutics within 2 weeks prior to start of study treatment. Antibody based agents within 4 weeks prior to start of study treatment. Mitomycin C or nitrosoureas within 6 weeks prior to start of study treatment.
* For participants who may get lorlatinib or encorafenib on study, history of interstitial lung disease
* For participants who may get binimetinib on study, history or current evidence of retinal vein occlusion (RVO) or concurrent neuromuscular disorder associated with elevated creatine kinase (CK)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2024-06-19 (Actual); Study Completion 2024-06-19 (Actual)

PRIMARY OUTCOMES:
Part 1 and Part 2- Number of participants with dose limiting toxicities (DLTs) | Cycle 1 (21 days)
  DLTs will be evaluated during the first cycle (21 days) as both a single agent or in combination with lorlatinib, encorafenib + cetuximab, or binimetinib. The number of DLTs will be used to determine the maximum tolerated dose (MTD)/recommended dose for further study
Part 1 and Part 2- Number of participants with treatment-emergent adverse events (AEs) | Baseline up to 30 days after last dose of study medication
  AEs as characterized by type, frequency, severity, timing, seriousness, and relationship to study therapy
Part 1 and Part 2 - Number of participants with clinically significant change from baseline in laboratory abnormalities | Baseline up to 30 days after last dose of study treatment
  Laboratory abnormalities as characterized by type, frequency, severity, and timing
Part 1 and Part 2 - Number of dose interruptions, dose modifications, and discontinuations due to AEs | Baseline up to 30 days after the last dose of study medication
  Incidence of dose interruptions, dose modifications, and discontinuations due to AEs
Part 3- Overall response | Baseline to up to 2 years
  Response will be evaluated via radiographical tumor assessments by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1)

SECONDARY OUTCOMES:
Part 1 and Part 2- Maximum plasma concentration (Cmax) of PF-07284892 and metabolite | Cycle 1 Day 1 (predose, 1, 2, 4, 6, 8 hours postdose); Cycle 1 Day 18 (predose, 1, 2, 4, 6, 8, 24, and 48 hours postdose); Cycle 2-6 Day 1 (predose and 2 hours postdose); Cycle 7-12 Day 1 predose; end of treatment (EOT)
  single dose (Cmax) and multiple dose (assuming steady state is achieved; Css,max) pharmacokinetic (PK) parameters
Part 1 and Part 2- Time to reach maximum plasma concentration (Tmax) of PF-07284892 and metabolite | Cycle 1 Day 1 (predose, 1, 2, 4, 6, 8 hours postdose); Cycle 1 Day 18 (predose, 1, 2, 4, 6, 8, 24, and 48 hours postdose); Cycle 2-6 Day 1 (predose and 2 hours postdose); Cycle 7-12 Day 1 predose; EOT
  Single dose (Tmax) and multiple dose (assuming steady state is achieved; Tss,max) pharmacokinetic parameters
Part 1 and Part 2- Area under the plasma concentration-time curve from time 0 to the last time point of quantifiable concentration (AUClast) of PF-07284892 and metabolite | Cycle 1 Day 1 (predose, 1, 2, 4, 6, 8 hours postdose); Cycle 1 Day 18 (predose, 1, 2, 4, 6, 8, 24, and 48 hours postdose); Cycle 2-6 Day 1 (predose and 2 hours postdose); Cycle 7-12 Day 1 predose; EOT
  Single dose PK parameter
Part 1 and Part 2- Area under the plasma concentration-time curve from time 0 to extrapolated to infinity (AUCinf) of PF-07284892 and metabolite | Cycle 1 Day 1 (predose, 1, 2, 4, 6, 8 hours postdose); Cycle 1 Day 18 (predose, 1, 2, 4, 6, 8, 24, and 48 hours postdose); Cycle 2-6 Day 1 (predose and 2 hours postdose); Cycle 7-12 Day 1 predose; EOT
  Single dose and multiple dose (assuming steady state is achieved) PK parameter
Part 1 and Part 2- Metabolite ratio of PF-07284892 and metabolite | Cycle 1 Day 1 (predose, 1, 2, 4, 6, 8 hours postdose); Cycle 1 Day 18 (predose, 1, 2, 4, 6, 8, 24, and 48 hours postdose); Cycle 2-6 Day 1 (predose and 2 hours postdose); Cycle 7-12 Day 1 predose; EOT
  Single dose PK parameter
Part 1 and Part 2- Area under the plasma concentration-time curve from 0 to 24 (AUC24) or 48 hours (AUC48) of PF-07284892 and metabolite | Cycle 1 Day 1 (predose, 1, 2, 4, 6, 8 hours postdose); Cycle 1 Day 18 (predose, 1, 2, 4, 6, 8, 24, and 48 hours postdose); Cycle 2-6 Day 1 (predose and 2 hours postdose); Cycle 7-12 Day 1 predose; EOT
  Multiple dose (assuming steady state is achieved) PK parameter
Part 1 and Part 2- Overall response | Baseline to up to 2 years
  Response will be evaluated via radiographical tumor assessments by RECIST v1.1
Part 2- Duration of Response (DOR) | Baseline to up to 2 years
  Time from the first documentation of objective response to the first documentation of objective progressive disease, relapse or to death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (19):
- United States (19):
  - Mayo Clinic in Arizona - Phoenix, Phoenix, Arizona
  - Mayo Clinic, Scottsdale, Arizona
  - California Cancer Associates for Research and Excellence, Encinitas, California
  - California Cancer Associates for Research and Excellence, San Marcos, California
  - University of Iowa, Iowa City, Iowa
  - Brigitte Harris Cancer Pavilion, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - START Midwest, Grand Rapids, Michigan
  - Henry Ford Medical Center - Columbus, Novi, Michigan
  - Mayo Clinic in Rochester, Minnesota, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Center David H Koch Center for Cancer Care, New York, New York
  - Memorial Sloan Kettering Cancer Center Rockefeller Outpatient Pavilion, New York, New York
  - Tennessee Oncology PLLC, Franklin, Tennessee
  - Tennessee Oncology, PLLC, Franklin, Tennessee
  - Sarah Cannon Research Institute- Pharmacy, Nashville, Tennessee
  - SCRI Oncology Partners, Nashville, Tennessee
  - Tennessee Oncology PLLC, Nashville, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4481001